CLINICAL TRIAL: NCT00389129
Title: Comparative Evaluation of Aspirin Resistance With Point-of-Care Testing - Danish Aspirin Resistance Trial (DANART) - Pilot Study
Brief Title: Danish Aspirin Resistance Trial - Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Danish Research Agency (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20060142
Record Dates: First submitted 2006-10-17; First posted 2006-10-18 (Estimated); Last update posted 2007-12-12 (Estimated); Status verified 2007-12

CONDITIONS: Drug Resistance
Keywords: Platelets; Aspirin Resistance; Platelet aggregation
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: acetylsalicylic acid

SUMMARY:
Despite treatment with aspirin a large number of patients suffer a myocardial infarction. It has been speculated that these patients might be "resistant" to aspirin, and studies have indicated that this phenomenon is related to a less favourable prognosis. At present, no international consensus exists on how to measure "aspirin resistance". The purpose of this study is to compare different methods for detecting "aspirin resistance". A classic but cumbersome way of evaluating platelet function will be compared to newer, easy-handling point-of-care tests. We hypothesize that one or more point-of-care tests will prove to be superior to the classic platelet function test in detecting aspirin resistance.

DETAILED DESCRIPTION:
Platelets play a major role in arterial thrombus formation - the cause of cardiovascular death, acute myocardial infarction and ischemic stroke and the number one killer in the Western World. Binding the COX enzyme platelet aggregation is inhibited by aspirin, and as prophylaxis against death, myocardial infarction and stroke aspirin is the most widely used drug worldwide. Low dose aspirin has been shown to improve outcome in patients with ischemic heart disease, but approximately 12% of these patients will suffer from a vascular event during a 2 year follow-up period despite aspirin therapy. It has been speculated that these patients might be "resistant" to the antiaggregatory effect of aspirin, and a diminished response to aspirin has been correlated with a less favourable outcome. However, at present no international consensus exists on how to measure "aspirin resistance".

Comparisons: The platelet aggregation in patients with ischemic heart disease on chronic, low dose aspirin is compared to platelet aggregation i healthy volunteers evaluated with different tests. The traditional way of evaluating platelet function, Platelet Aggregometry a.m. Born, will be compared to 3 point-of-care tests (VerifyNow, PFA-100 and Multiplate Whole Blood Aggregometer) and to urin- and serum thromboxane metabolites as a measure of COX inhibition.

ELIGIBILITY:
Inclusion Criteria:

* ischemic heart disease verified with a coronary angiogram
* treatment with 75 mg aspirin once daily

Exclusion Criteria:

* ischemic vascular event within the previous 12 months
* percutaneous coronary intervention or coronary artery by-pass grafting within the previous 12 months
* treatment with NSAID, clopidogrel, ticlopidine, dipyridamole, warfarin or any other drug affecting platelet aggregation
* platelet count < 120 x 10^9/l
* not able to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2006-11; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Platelet aggregation (as determined by 3 point-of-care tests and by serum-thromboxane A2 + urine 11-dehydro thromboxane B2) is measured once daily for 4 days after one week of treatment with aspirin 75 mg/day

CONTACTS AND LOCATIONS:
Overall Officials: Steen D Kristensen, MD, DMSc, Study Director — Department of Cardiology, Skejby Sygehus, Aarhus University Hospital, 8200 Aarhus N, DK - Denmark; Erik L Grove, MD, Principal Investigator — Department of Cardiology, Skejby Sygehus, Aarhus University Hospital, 8200 Aarhus N, DK - Denmark
Locations (1):
- Department of Cardiology, Skejby Sygehus, Aarhus University Hospital, Aarhus, Denmark